CLINICAL TRIAL: NCT06771895
Title: Post Intensive Care Optimization Through Lifestyle Intervention
Acronym: PICOLI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 24-059
Record Dates: First submitted 2024-12-10; First posted 2025-01-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: ICU Survivor; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: This study can be defined as a single-group (uncontrolled) clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Combined exercise and nutritional intervention

INTERVENTIONS:
Behavioral: Combined exercise and nutritional intervention — The intervention consists of a combined exercise and nutritional intervention. All subjects will perform 20 weeks of supervised resistance and endurance type exercise training 2 to 3 days per week. The dietary intervention aims to attain a diet that comprises sufficient protein and is otherwise in line with the Dutch Healthy Diet guidelines. In support, subjects will consume a daily high protein multi-nutrient supplement which will be ingested pre-sleep. There will be an additional supplement intake moment following each training session.

SUMMARY:
The quality of the intensive care unit (ICU) has been steadily improving over the years. Although improvements in the acute treatment of critically ill patients have been made, a large number of ICU survivors suffer from severe physical, cognitive and mental health problems persisting months to years after leaving the ICU. Physical impairments occur the most and can be very severe, greatly affecting activities in daily life and subsequently the perceived quality of life of ICU survivors. Although there is an increased awareness of long-term complaints following ICU stay, there is currently a knowledge gap on how to enhance the recovery of ICU survivors 6 to 12 months post-ICU discharge. The overall objective of the current study is to establish the extent of health and functional improvements that can be obtained with an optimized, combined exercise and nutritional intervention in ICU survivors 6 to 12 months post-ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Minimum ICU length of stay of 5 days and/or mechanically ventilated for a minimum of 2 days
* Persistent physical complaints
* Community-dwelling, living independently (non-assisted)
* Mentally competent with a Mini-Mental State Examination (MMSE) score of ≥24
* Willing to participate in a 20-week multimodal lifestyle intervention

Exclusion Criteria:

* Any medical condition that may interfere with the safety of the subjects during exercise or any condition that interferes with assessment of the outcome parameters, in the investigators' judgement in consultation with the responsible physician or treating physician/specialist. In case of a contra-indication for MRI (e.g., a pacemaker), subjects will be excluded from this measurement but not necessarily from the study.
* Any medical condition or circumstance where supplementation with the nutritional supplement is potentially contra-indicated.
* Known allergy to any of the ingredients present in the nutritional supplement.
* Simultaneous use of other nutritional supplements during the study period (i.e., unwillingness to stop for the duration of the study).
* Current participation in other scientific research that conflicts with this study (e.g. intervention studies or weight management studies).
* No permission to request information from the general practitioner/treating specialist(s) about medical history, medication use.

  * Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by a VO2-peak test on ergometer
Muscle strength | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by 1-RM max testing
Muscle mass | At baseline (week 0) and at the end of the intervention (week 22)
  as measured by whole-body MRI

SECONDARY OUTCOMES:
Body fat composition | At baseline (week 0) and at the end of the intervention (week 22)
  as measured by whole-body MRI
Body lean mass composition | At baseline (week 0) and at the end of the intervention (week 22)
  as measured by whole-body MRI
Metabolic health | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  by assessing nutritional status, lipid profile, inflammatory profile, fasting glucose and insulin in plasma and serum samples
Gut health | In week 1, week 4 and week 21 of the intervention
  by assessing intestinal microbiota composition, diversity and taxa abundance, functional capacity of the intestinal microbiota and metabolomics in feces samples
Brain health (cognitive function) | At baseline (week 0) and at the end of the intervention (week 22)
  as measured by the Cambridge Neuropsychological Test Automated Battery
Step count | In week 1, week 11 and week 21 of the intervention
  as measured by accelerometry
Age | At baseline (week 0)
  as measured using a questionnaire
Body mass | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by a scale
Height | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by a stadiometer
Body Mass Index | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as calculated from height and body mass
Waist circumference | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by measuring tape
Systolic and diastolic blood pressure | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured using an automated device
Handgrip strength | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by a dynamometer
Functional capacity | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the 6-Minute Walk Test
Physical function | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Short Physical Performance Battery
Muscle fiber size | At baseline (week 0) and at the end of the intervention (week 22)
  as determined by immunofluorescence staining of muscle biopsy of vastus lateralis (optional)
Myonuclei quantity | At baseline (week 0) and at the end of the intervention (week 22)
  as determined by immunofluorescence staining of muscle biopsy of vastus lateralis (optional)
Proportion (%) of muscle fiber types (type I and type II) | At baseline (week 0) and at the end of the intervention (week 22)
  as determined by immunofluorescence staining of muscle biopsy of vastus lateralis (optional)
Frailty | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Clinical Frailty Scale
Quality of Life | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Short Form 36 Health Survey v2 and EuroQol-5 Dimensions-5 Levels questionnaires
Mental health | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Hospital Anxiety & Depression Scale
Sleep quality | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Pittsburgh Sleep Quality Index
Supplement tolerance | At baseline (week 0), midline (week 11) and at the end of the intervention (week 22)
  as measured by the Gastrointestinal Symptom Rating Scale
Intestinal transit rate | In week 1, week 4 and week 21 of the intervention
  as measured by the Bristol Stool Scale
Dietary protein intake | In week 1, week 4 and week 21 of the intervention
  as measured by dietary diaries
Dietary carbohydrate intake | In week 1, week 4 and week 21 of the intervention
  as measured by dietary diaries
Dietary fat intake | In week 1, week 4 and week 21 of the intervention
  as measured by dietary diaries

CONTACTS AND LOCATIONS:
Overall Officials: Lex B Verdijk, Dr., Principal Investigator — Maastricht University; Luc JC van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Center+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined